CLINICAL TRIAL: NCT03316794
Title: An Open-Label Study of SC-005 in Subjects With Triple Negative Breast Cancer (TNBC)
Brief Title: A Study of SC-005 in Subjects With Triple Negative Breast Cancer (TNBC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-735
Record Dates: First submitted 2017-10-18; First posted 2017-10-20 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
Keywords: Triple Negative Breast Cancer; Cancer; Breast Cancer; Maximum tolerated dose (MTD); Pharmacokinetics
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SC-005 (Experimental): SC-005 intravenous (IV) (various doses and dose regimens)
  Interventions: Drug: SC-005

INTERVENTIONS:
Drug: SC-005 — intravenous

SUMMARY:
This is a multicenter, open-label study in participants with triple negative breast cancer (TNBC) to study the safety, tolerability, pharmacokinetics and preliminary efficacy of SC-005. This study consists of 2 parts: Part A (dose regimen finding) followed by Part B (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced TNBC that is relapsed, refractory, or progressive and not eligible for another standard therapy that would confer clinical benefit to the subject.

  * Advanced disease is defined as metastatic disease or locally advanced disease that is not amenable to surgery or radiotherapy with curative intent
  * TNBC is defined as:
* <1% staining by immunohistochemistry (IHC) for estrogen (ER) and progesterone (PR) receptors, 0 or 1+ IHC for human epidermal growth factor receptor 2 (HER2), OR
* Negative for HER2 amplification by in situ hybridization (ISH) for 2+ IHC disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Any significant medical condition including any suggested by Screening laboratory findings that, in the opinion of the Investigator or Sponsor, may place the subject at undue risk from the study.
* Has ECG abnormalities that make QT interval corrected (QTc) evaluation difficult (e.g., severe morphologic abnormalities).
* Prior exposure to a pyrrolobenzodiazepine or indolino-benzodiazepine based drug, or known hypersensitivity or contraindication to SC-005 or excipient contained in the drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | Minimum 21 days
  DLTs graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
QTcF Change from Baseline | Up to approximately 9 weeks
  QT interval measurement corrected by Fridericia's formula (QTcF)
Area Under the Plasma Concentration-time Curve (AUC) | Up to approximately 9 weeks
  Area under the plasma concentration-time curve (AUC) of SC-005.
Clinical benefit rate (CBR) | Up to approximately 4 years
  CBR is defined as the proportion of participants with an objective response or stable disease (CR+PR +SD).
Maximum plasma concentration observed (Cmax) | Up to approximately 9 weeks
  Maximum plasma concentration observed (Cmax) of SC-005
Overall Survival (OS) | Up to approximately 4 years
  OS is defined as the time from the participant's first dose date to death due to any cause.
Observed Plasma Concentrations at Trough | Up to approximately 9 weeks
  Observed plasma concentrations at trough of SC-005.
Duration of Clinical Benefit (DOCB) | Up to approximately 4 years
  DOCB is defined as the time from the participant's initial observation of clinical benefit (CR or PR or stable disease [SD]) to PD or death due to any cause, whichever occurs first.
Objective Response Rate (ORR)Up to approximately 4 years | Up to approximately 4 years
  Objective response rate is defined as the proportion of participants with complete response (CR) or partial response (PR) based on RECIST version 1.1.
Time of Cmax (Tmax) | Up to approximately 9 weeks
  Time of Cmax (Tmax) of SC-005.
Progression Free Survival (PFS) | Up to approximately 4 years
  PFS time is defined as the time from the participant's first dose of study drug (Day 1) to either the participant's disease progression or death due to any cause.
Duration of Response (DOR) | Up to approximately 4 years
  DOR is defined as the time from the participants initial objective response (CR or PR) to disease progression (PD) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (8):
- United States (8):
  - University of Chicago /ID# 169231, Chicago, Illinois
  - Washington University School /ID# 169177, St Louis, Missouri
  - Memorial Sloan Kettering /ID# 201016, New York, New York
  - Gabrail Cancer Center Research /ID# 168756, Canton, Ohio
  - Oklahoma University /ID# 200937, Oklahoma City, Oklahoma
  - Tennessee Oncology-Sarah Cannon Research Institute /ID# 169233, Nashville, Tennessee
  - Baylor University /ID# 169860, Houston, Texas
  - MD Anderson Cancer Center /ID# 169232, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided